CLINICAL TRIAL: NCT00816114
Title: Chart Review Study of Chronic Myelogenous Leukemia (CML) Patients Treated With Imatinib Outside of a Clinical Trial
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: RCR05-0444; NCI-2021-13238 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2008-12-30; First posted 2008-12-31 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Imatinib; Gleevec; Chronic Myelogenous Leukemia; CML
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Myelogenous Leukemia: All CML patients in any phase of the disease that received imatinib treatment outside of MDACC clinical trials and has had at least one MDACC clinic visit.
  Interventions: Other: Chart Review

INTERVENTIONS:
Other: Chart Review — Investigator review of MDACC CML patient charts.

SUMMARY:
In this study researchers propose to do a chart review of all patients that are treated outside of a clinical trial with imatinib, dasatinib, nilotinib, or any other tyrosine kinase inhibitor that becomes FDA approved for the managements of CML that come to MDACC for a second opinion. This is an important population of patients that differs in their management from patients treated in clinical trials for several reasons including but not limited to:

1. It represents a very large patient population receiving standard-dose therapy with TKI. We estimate that we have evaluated over 300 patients that fall in this category.
2. The follow-up for patients in the largest trial using standard-dose imatinib (the IRIS trial, with 553 patients in treated with imatinib) has been limited after the first 12 months. For example, the rate of molecular responses after the first 12 months of therapy was not obtained as samples stopped being collected at that time point.
3. Registration studies for dasatinib and nilotinib have similar limitations with limited follow-up and available information coming only from databases from the sponsors to which there is limited access to investigate dosing, chronic toxicities, second malignancies and other important aspects of therapy.
4. Patients who are or become pregnant during therapy with TKI have not been eligible for clinical trials with TKI or had to be taken off study. Thus, there is no information on the effect of TKI on imatinib on pregnancy and conception. We have followed several such patients at MDACC.
5. This is a patient population that follows therapy mostly as directed by their local oncologists. This is frequently less stringently adhered to the recommended guidelines for TKI therapy, with more frequent treatment interruptions, and frequently using suboptimal doses of imatinib (i.e., less than 300mg daily). The effect of these treatment interruptions and suboptimal dosing on response and development of resistance is unclear.

Researchers plan to conduct a chart review of these patients to study their treatment course before their initial evaluation at MDACC, and between and during visits to MDACC.

DETAILED DESCRIPTION:
PATIENT POPULATION:

All patients with CML in any phase of the disease (chronic, accelerated or blast phase) that has received treatment with any tyrosine kinase inhibitor (eg, imatinib, dasatinib, nilotinib) regardless of prior treatment history that has had at least one clinic visit at MDACC will be eligible.

STUDY PLAN:

The following information will be collected:

* Demographic information including age, gender, ethnicity, education, and work history.
* All laboratory values obtained at MDACC or other institutions, including CBC, blood chemistries, electrolytes, bone marrow aspirations and biopsies, cytogenetic analyses, mutation analysis, FISH, and PCR, and other tests obtained during regular care of these patients.
* Treatment history including starting and stopping dates, doses, treatment interruptions, dose changes and reasons for dose modifications.
* Information about toxicity including type, grade, dates of onset and resolution, interventions to manage toxicity, and sequelae.
* Information regarding pregnancy or conception during imatinib therapy for both male and female patients, including dates of pregnancy, outcome of pregnancy, interventions during pregnancy, management of CML during pregnancy, complications during pregnancy, status of the product, condition of the born child, and information on lactation.
* This information will be reviewed from the documents received as part of the routine communication with the local oncologist or from the studies obtained at MDACC.
* There will be no treatment changes or recommendations as a result of this study. This study will be strictly limited to review of charts. Patients will continue their treatment as recommended by their local oncologist and treating physician at MDACC.
* These results will be compared to similar patients treated with imatinib in the context of clinical trials both from published literature and from other studies conducted at MDACC. The efficacy, safety and prognostic markers will be compared.
* We will review data from July 1, 1998 to August 1, 2019.

SAMPLE SIZE:

Approximately 3000 charts will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

All patients with CML in any phase of the disease (chronic, accelerated or blast phase) that has received treatment with any FDA-approved tyrosine kinase inhibitor (eg, imatinib, dasatinib, nilotinib) not on an MDACC clinical trial regardless of prior treatment history that has had at least one clinic visit at MDACC will be eligible.

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MDACC CML patients (July 1, 1998 to September 1, 2017) in any disease phase (chronic, accelerated or blast phase) that received imatinib treatment outside an MDACC clinical trial prior to a MCACC clinic visit.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2005-06-08 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
CML Patient Response to standard dose imatinib treated outside clinical trial setting | June 2012

SECONDARY OUTCOMES:
Number of chromosomal abnormalities incidences in Ph-negative metaphases associated with imatinib treatment in CML patients treated with standard dose outside clinical trial setting | June 2012
Outcome of conception + pregnancy during imatinib treatment in CML patients | June 2012

CONTACTS AND LOCATIONS:
Overall Officials: Koji Sasaki, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Assi R, Kantarjian H, Keating M, Pemmaraju N, Verstovsek S, Garcia-Manero G, Ravandi F, Borthakur G, Dahl J, Jabbour E, Cortes JE. Management of chronic myeloid leukemia during pregnancy among patients treated with a tyrosine kinase inhibitor: a single-Center experience. Leuk Lymphoma. 2021 Apr;62(4):909-917. doi: 10.1080/10428194.2020.1849672. Epub 2020 Dec 7. PMID 33283580
- See also: MD Anderson Cancer Center Website — http://mdanderson.org